CLINICAL TRIAL: NCT03129243
Title: Relation of Sperm DNA Damage to Intracytoplasmic Sperm Injection Outcome in Couples With Male Infertility
Brief Title: Sperm DNA Damage to Intracytoplasmic Sperm Injection Outcome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: ICSI
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sperm DNA integrity by flow cytometry — flowcytometric test where sperm DNA breaks are evaluated indirectly through the DNA denaturability. The assay measures the susceptibility of sperm DNA to acid-induced DNA denaturation in situ, followed by staining with the fluorescence dye acridine orange. By using a flow cytometer 5.000-10.000 sperm can be analyzed within few seconds and thus provide a less subjective result compared to the World health organization analysis where only 1-300 cells are analyzed.

SUMMARY:
In the current era of assisted reproductive techniques where technology can help overcome defects in sperm function, the value of semen analysis has become even more inaccurate. Initial reports of intracytoplasmic sperm injection revealed its ability to bypass the natural selection process and enable men with severely impaired semen parameters to achieve both clinical pregnancy and live birth

ELIGIBILITY:
Inclusion Criteria:

1. Infertile male patients with abnormal semen parameters.
2. Normal female partner aged <38 years.

Exclusion Criteria:

1. Female patients with obvious infertility factor.
2. Male patients with azoospermia.
3. Male patients with systemic diseases.
4. Male patients receiving cytotoxic therapy.
5. Male patients with genital pathology as cryptorchidism.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include all infertile couples undergoing intracytoplasmic sperm injection in The Department of Dermatology and Andrology with assisted reproductive unit at women's health hospital, Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided